CLINICAL TRIAL: NCT05513482
Title: Prospective Evaluation of Diaphragm Kinetics With Tissue Doppler Imaging in Patients Undergoing Atrial Fibrillation Ablation With Cryoballoon
Brief Title: Ultrasonography Evaluation of Diaphragm Kinetics in Patients Undergoing Atrial Fibrillation Ablation With Cryoballoon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz Mutlu, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 2022/449352
Record Dates: First submitted 2022-08-11; First posted 2022-08-24 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation; Phrenic Nerve Paralysis
Keywords: Pulmonary vein isolation; Atrial fibrillation ablation; Arrhythmia; Phrenic nerve; Tissue doppler imaging; Diaphragm kinetics
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cryoballoon pulmonary vein isolation for atrial fibrillation ablation: Diaphragmatic kinetics of participants before and after pulmonary vein isolation will be evaluated with the Tissue Doppler and M Mode Imaging.
  Interventions: Diagnostic Test: Tissue Doppler Imaging; Diagnostic Test: M Mode Imaging

INTERVENTIONS:
Diagnostic Test: Tissue Doppler Imaging — With tissue Doppler ultrasonography (TDI), the maximum contraction rate of the diaphragm, maximum relaxation rate, and integral against time will be examined.
  Other Names: GE Vivid T8 Ultrasonography System
Diagnostic Test: M Mode Imaging — Diaphragm displacement during inspiration and expiration will be measured with M mode imaging
  Other Names: GE Vivid T8 Ultrasonography System

SUMMARY:
The purpose of this study to assess the diaphragm kinetics with Tissue Doppler Imaging in patients undergoing atrial fibrillation ablation with cryoballoon

DETAILED DESCRIPTION:
This study is designed to evaluate the diaphragm kinetics with ultrasonography parameters in patients who underwent pulmonary vein isolation (PVI) for atrial fibrillation (AF) by Cryoballoon. Due to the proximity of the pulmonary veins to the phrenic nerve, phrenic nerve paralysis can be seen rarely during the procedure. In contemporary practice, phrenic nerve damage is detected by visual monitoring of diaphragm movement as a result of pacing with high output by placing the intracardiac stimulation catheter at the level of the superior vena cava. However, subclinical nerve damage may be critical regarding respiratory functions, especially in patients with comorbidities. It has been shown in the literature that the evaluation of diaphragm kinetics with Tissue Doppler Imaging (TDI) can be used in effective ventilation monitoring and weaning. However, this technique has not been used in patients who have previously undergone cryoballoon therapy. It is aimed to investigate the positive or negative effects on diaphragm kinetics, as a very cost-effective and rapidly accessible technique, with the help of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for AF ablation with a cryoballoon
* ≥18 years old
* Patients with interpretable diaphragm ultrasound before the operation
* Patients giving informed consent

Exclusion Criteria:

* Patients who did not give consent
* Patients with phrenic nerve palsy
* Morbid obesity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population will consist of patients who are planned for AF ablation with the cryobaloon, whose preoperative ultrasonography can be interpreted and who gave their consent.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-23 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Detection of subclinical phrenic nerve injury with changes in diaphragm kinetics, before and after the procedure | Preoperative baseline and postoperative first hour
  Unlike the traditional method, diaphragm Tissue Doppler imaging (TDI) will be used to diagnose phrenic nerve injury in patients during cryoballoon ablation. This method aims to detect the damages that may have occurred even though no visible damage has occurred. The peak contraction velocity (PCV) that has been found to be effective on weaning success will be used in TDI. The literature shows that the PCV measured by TDI in healthy humans is 1.32 ⨦ 0.39 cm/sec. Based on this, the patient's baseline and post-procedure PCVs will be compared.

SECONDARY OUTCOMES:
The effect of subclinical diaphragm damage on morbidity | Preoperative baseline and postoperative 24 hours
  Side effects that may occur as a consequence of these will be observed in patients with subclinical diaphragm injury.

CONTACTS AND LOCATIONS:
Overall Officials: Kivanc Yalin, Assoc Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505
- [Result] Soilemezi E, Savvidou S, Sotiriou P, Smyrniotis D, Tsagourias M, Matamis D. Tissue Doppler Imaging of the Diaphragm in Healthy Subjects and Critically Ill Patients. Am J Respir Crit Care Med. 2020 Oct 1;202(7):1005-1012. doi: 10.1164/rccm.201912-2341OC. PMID 32614246
- [Result] Cammarota G, Boniolo E, Santangelo E, De Vita N, Verdina F, Crudo S, Sguazzotti I, Perucca R, Messina A, Zanoni M, Azzolina D, Navalesi P, Longhini F, Vetrugno L, Bignami E, Della Corte F, Tarquini R, De Robertis E, Vaschetto R. Diaphragmatic Kinetics Assessment by Tissue Doppler Imaging and Extubation Outcome. Respir Care. 2021 Jun;66(6):983-993. doi: 10.4187/respcare.08702. Epub 2021 Apr 27. PMID 33906957
- [Result] Tokuda M, Yamashita S, Sato H, Oseto H, Ikewaki H, Yokoyama M, Isogai R, Tokutake KI, Yokoyama KI, Kato M, Narui R, Tanigawa SI, Matsuo S, Yoshimura M, Yamane T. Long-term course of phrenic nerve injury after cryoballoon ablation of atrial fibrillation. Sci Rep. 2021 Mar 18;11(1):6226. doi: 10.1038/s41598-021-85618-3. PMID 33737633